CLINICAL TRIAL: NCT00003970
Title: A Phase I Clinical Trial to Investigate the Correlation Between UGT1A1 Genotype and Irinotecan (CPT-11) Pharmacokinetics and Toxicity in Cancer Patients
Brief Title: Genetic Testing Plus Irinotecan in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02304; 9531; U01CA069852 (NIH); CDR0000067173 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Irinotecan

ARMS (1):
- Treatment (irinotecan hydrochloride) (Experimental): Patients receive irinotecan IV over 90 minutes once every 3 weeks. Treatment continues for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
Phase I trial to study genetic testing and the effectiveness of irinotecan in treating patients who have solid tumors and lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Genetic testing for a specific enzyme may help doctors determine whether side effects from or response to chemotherapy are related to a person's genetic makeup

DETAILED DESCRIPTION:
OBJECTIVES:

I. Classify patients with solid tumors or lymphoma according to UGT1A1 promoter (TATA box) and coding region (Gly71Arg) mutation, and CYP3A4 promoter (G to A) polymorphisms.

II. Identify UGT1A1 enzyme glucuronidator and irinotecan oxidizer phenotypes in these patients and determine the correlation between the two metabolic reactions in vivo.

III. Determine the relationship between UGT1A1 genotype (promoter and/or coding region mutation) and CYP3A4 promoter genotype vs gastrointestinal or bone marrow toxicity, and pharmacokinetics of irinotecan in these patients.

IV. Determine the pharmacokinetics of irinotecan in these patients.

OUTLINE: Patients are genotyped for UGT1A1 enzyme and classified as "Gilbert's" (7/7), "heterozygotes" (6/7), and "homozygotes for allele 6" (6/6). The DNA is analyzed for the UGT1A1 coding region mutation (Gly71Arg) and CYP3A4 promoter polymorphism. Patients are also examined for glucuronidator ratio of SN-38, the active metabolite of irinotecan, and classified as "low/slow" (very low or zero SN-38G/SN-38 ratio), "intermediate" (less than 50% normal ratio), or "normal".

Patients receive irinotecan IV over 90 minutes once every 3 weeks. Treatment continues for at least 2 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven solid tumor or lymphoma

  * Responded to irinotecan OR no existing curative therapy
* No leukemia
* Measurable or evaluable disease
* Performance status - Karnofsky 70-100%
* WBC at least 3500/mm^3
* Absolute neutrophil count at least 1500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* SGOT/SGPT less than 5 times upper limit of normal (unless due to disease)
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No inflammatory bowel disease requiring therapy
* No chronic diarrhea syndrome or paralytic ileus
* At least 2 weeks since prior colony stimulating factor
* At least 4 weeks since prior biologic therapy
* No concurrent biologic therapy
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* At least 4 weeks since prior radiotherapy to greater than 25% of bone marrow
* No concurrent palliative radiotherapy
* No prior transplant
* No concurrent substrates of UGT1A1 enzyme
* No concurrent inducers or inhibitors of UGT1A1 enzyme activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1999-01; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Grade 3-4 diarrhea | Up to 4 years
  A Cochran-Armitage test for trend will be used to determine whether there is a linear trend in the proportion of patients within each genotype experiencing grade 3-4 diarrhea. Similarly, trend analysis will be performed to determine if there is a linear trend in the proportion of patients within each phenotype experiencing grade 3-4 myelosuppression. Genotype (3 ordered levels) will be modeled as a function of metabolic ratios and biliary index to determine whether these are independent.

SECONDARY OUTCOMES:
Genotype | Up to 4 years
  A chi-squared test will be used to determine whether genotype and phenotype are independent.
Phenotype | Up to 4 years
  A chi-squared test will be used to determine whether genotype and phenotype are independent. Modeled as a function of metabolic ratios and biliary index.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States